CLINICAL TRIAL: NCT05399446
Title: Multi-site Trial of a Virtually Delivered Eating Disorder Prevention Program for Young People with Type 1 Diabetes
Brief Title: Multi-Site Eating Disorder Prevention Program for Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of Minnesota (Other); Joslin Diabetes Center (Other); Stanford University (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Line Wisting, Researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 65953
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes; Eating Disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The assessor completing the interview at each follow-up assessment following completion of the intervention will be blinded to the condition the participant was in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Body Project (Experimental)
  Interventions: Behavioral: Diabetes Body Project
- Educational Group (Active Comparator)
  Interventions: Behavioral: Educational Group

INTERVENTIONS:
Behavioral: Diabetes Body Project — The Diabetes Body Project (DBP) is an adapted version of the Body Project Prevention program designed specifically for individuals with Type 1 Diabetes. DBP consists of six weekly, one-hour long sessions. Group participants complete the exercises from the original Body Project and also new diabetes-specific content, drawn from Olmsted et al. (2002) that is delivered in a dissonance-based interactive format with Socratic questions from group leaders encourage participants to generate their own answers.
  Arms: Diabetes Body Project
Behavioral: Educational Group — We selected a T1D management/Eating disorder psychoeducational comparison condition to control for expectancy effects and demand characteristics. To match the Diabetes Body Project, the educational lectures will be delivered in 6 1-hour blocks. Topics include basic information about the various EDs, complications of ED behaviors, diabetes and body image, effects of dieting on blood glucose, and the risk of complications.
  Arms: Educational Group

SUMMARY:
This study aims to test the effectiveness of an evidence-based eating-disorder prevention program specifically targeted for individuals with Type 1 Diabetes (T1D) compared to an educational control group. The Diabetes Body Project (DBP), is an adaptation of the Body Project which is the only eating disorder prevention program to have repeatedly produced effects when evaluated by independent researchers, produced stronger effects than credible alternative interventions, and affected objective outcomes. DBP has been adapted slightly for individuals with T1D who are at ultra-high risk for eating disorders. The study aims to test the effectiveness of the DBP of reducing body image concerns and reducing eating pathology and improving glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 14-35
2. diagnosis of Type 1 Diabetes of at least 1 year
3. using insulin
4. experiencing at least some level of body image concerns

Exclusion Criteria:

1. not between the ages of 14-35
2. does not have access to wifi (will need for the virtual groups)
3. Type 1 Diabetes diagnosis of less than 1 year
4. does not live in the same time zone of Stanford (helps in coordinating groups)
5. hospitalized for eating disorder treatment in the past year
6. had eating-disorder related Diabetic Ketoacidosis (DKA) in the past year
7. not using insulin
8. not experiencing any level of body image concerns
9. Unwilling to be video-recorded if assigned to Diabetes Body Project
10. restricted proficiency in language that groups will be conducted in (dependent on location), and pervasive developmental, cognitive, or psychiatric limitations that compromise participation in the intervention sessions and study.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Groups are single-gendered. Most participants (280) will be female-identifying. Each site is also going to recruit 1 group (about 6 individuals) of male-identifying individuals as to pilot the intervention with men. In total, there will be about 30 male-identifying individuals for a total sample of 310.
Enrollment: 280 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change over time in Ideal Body Beliefs | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Assessed with the 8-item Ideal-Body Stereotype Scale-Revised (Stice et al., 2017) which measures pursuit of the thin ideal. Each item is scored on a scale of 1 = strongly disagree to 5 = strongly agree. Higher scores indicate greater belief in the thin-deal.
Change over time in Body Dissatisfaction | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Assessed with the 10-item Body Dissatisfaction Scale (BDI; Berscheid et al., 2973) which assesses dissatisfaction with various body parts. Each item is scored on a scale of 1 = extremely dissatisfied to 5 = extremely satisfied. Lower scores indicate greater body dissatisfaction.
Change over time in Diabetes-Specific Eating Pathology | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Assessed with the 16-item Diabetes Eating Problem Survey-Revised (DEPS-R; Markowitz et al,.2010). Each item is assessed on a scale of 0 = Never to 5= Always. Higher scores indicate greater eating pathology specific to individuals with Type 1 Diabetes such as purposefully not taking enough insulin.
Change in Eating Disorder Symptoms | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Participants will complete a diagnostic interview that is administered by a trained research assistant. We will be using the Eating Disorder Diagnostic Interview (EDDI). Scores are not reported on a scale. The research assistant who conducts the diagnostic interview at post-test and 3-month follow-up will be blinded to the person's condition.

SECONDARY OUTCOMES:
Change in Glycemic Control | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Objectively assessed HbA1c (at clinic or by a self-test kit)
Change in Time-In-Range (TIR) | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  TIR past 14 days, screen shot of device. Time-Above-Range (TAR) and Time-Below-Range (TBR) are also recorded
Change in Health Care Utilization | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  service utilization will be assessed with an adapted version of the Patterns of Help Seeking Behavior Scale (Lane & Addis, 2005). Participants in both conditions will be asked to report frequency of care the past year for physical, mental health, eating, and weight problem
Change over time in Diabetes-Specific Distress | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Assessed with the 20-item Problem Areas In Diabetes scale (PAID) which measures distress related to diabetes. High scores indicate greater distress that are related to living with Type 1 Diabetes
Change over time in Diabetes-Related Quality of Life | pre intervention obtained on intake, immediately post intervention, 6 months, 1-year, and 2-years after the conclusion of the intervention]
  Assessed with the adolescent version (23 items) (Hilliard et al., 2020)and young adult version (27-items) of Type 1 Diabetes and Life (T1DAL) measures (Hilliard et al., 2021)assess diabetes specific health-related quality of life among participants with T1D. Total scores are transformed to a 0-100 scale and enables comparison of scores across age ranges. Higher scores indicate greater distress.

CONTACTS AND LOCATIONS:
Overall Officials: Line Wisting, PhD, Principal Investigator — Oslo University Hospital; Eric Stice, PhD, Principal Investigator — Stanford University; Elena Toschi, MD, Principal Investigator — Joslin Diabetes Center; Maartje de Wit, PhD, Principal Investigator — Amsterdam Medical University Centers
Locations (4):
- United States (2):
  - Stanford University, Stanford, California
  - Joslin Diabetes Center, Boston, Massachusetts
- Amsterdam Medical University Center, Amsterdam, Netherlands
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haugvik S, Hennekes M, Stice E, de Wit M, Toschi E, Wisting L. The diabetes body project: Study protocol of a multi-site trial of a virtually delivered eating disorder prevention program for young women with type 1 diabetes. Diabet Med. 2024 Sep;41(9):e15334. doi: 10.1111/dme.15334. Epub 2024 May 9. PMID 38721639